CLINICAL TRIAL: NCT03368131
Title: A Prospective Study of Concurrent Neoadjuvant Chemoradiotherapy Plus Trastuzumab for Siewert II ，III of HER-2 Positive Adenocarcinoma at Gastroesophageal Junction
Brief Title: Concurrent Neoadjuvant Chemoradiotherapy Plus Trastuzumab in the Treatment of Siewert II ，III of Human Epidermal Growth Factor Receptor-2(HER-2) Positive Gastroesophageal Junction Adenocarcinoma： A Randomized, Controlled Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alien Crafe 0005
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Trastuzumab; Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab XELOX and radiotherapy (Experimental): Trastuzumab is intravenously administered with the loading dose of 8 mg/kg followed by maintenance dose of 6mg/kg in day 1 of each cycle. XELOX：Capecitabine 825~1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45 Gray (unit)Gy/25f （1.8Gy/f/d，5 f/w）
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy
- XELOX and radiotherapy (Active Comparator): Capecitabine：825~1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45Gy/25f （1.8Gy/f/d，5 f/w）
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Trastuzumab — intravenously administered with the loading dose of 8 mg/kg followed by maintenance dose of 6mg/kg in day 1 of each cycle
  Arms: Trastuzumab XELOX and radiotherapy
Drug: Capecitabine — 825~1000mg/m2 bid d1-14
Drug: Oxaliplatin — 130 mg/m2 Ivgtt d1 q3w
Radiation: Radiotherapy — 45 Gray (unit) Gy/25f （1.8Gy/f/d，5 f/w）

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive concurrent neoadjuvant chemoradiotherapy for Siewert II ，III of locally advanced HER-2 Positive adenocarcinoma at gastroesophageal junction

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 60 years old (man or female);
* confirmed to Siewert II , III of locally advanced adenocarcinoma at gastroesophageal junction. The her-2 positive was detected by immunohistochemistry or Fluorescence in SituHybridization(FISH);
* Patients with Stage for Ⅲ by Endorectal Ultrasonography( EUS), Computed Tomography(CT) (or Positron Emission Tomography(PET )-CT) and laparoscopic (According to the eighth edition of American Joint Committee on Cancer (AJCC) );
* Patients are diagnosed as potentially resectable by multidisciplinary team, no surgical contraindications, and expected to be surgical resection;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Major organ function has to meet the following criteria:

HB≥80g/L; ANC≥1.5×109/L; PLT≥90×109/L; Alanine Transaminase (ALT) and Aspartate Transaminase(AST)≤2.5×ULN, but<≤5×ULN if the transferase elevation is due to liver metastases； Total Bilirubin(TBIL)<1.5×ULN； Serum creatinine ≤1.5×ULN;Serum albumin ≥ 30g / L

* Life expectancy greater than or equal to 6 months;
* Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

* Allergic to trastuzumab, capecitabine and oxaliplatin;
* severe diseases such as liver and kidney，myocardial infarction, symptomatic congestive heart failure (CHF) (NYHA classes II-IV), unstable angina or serious cardiac arrhythmia，which affect the situation of chemotherapy or surgery
* A variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc);
* Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (+ +); Has melena and hematemesis in two months;
* Coagulant function abnormality (International Normalized Ratio(INR) > 1.5 ULN, Activated Partial Thromboplastin Time(APTT ) > 1.5 ULN), with bleeding tendency;
* Pregnant or lactating women;
* Patients with other malignant tumors within 5 years (except for curable skin basal cell carcinoma and cervical carcinoma in situ);
* History of psychiatric drugs abuse and can't quit or patients with mental disorders;
* Less than 4 weeks from the last clinical trial;
* The researchers think inappropriate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response rate(pCR) | within 3 weeks after surgery
  The lesion disappeared completely by pathology

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Baseline to measured date of death from any cause
Disease-free survival(DFS) | 3 years
  Baseline to measured date of recurrence or death from any cause
Disease Control Rate (DCR) | 3 years
  Percentage of participants who achieved a best overall response of CR or PR or Stable Disease (SD).
Percentage of Participants With Objective Response According to Modified Response Evaluation Criteria In Solid Tumors(mRECIST) v1.1 | within 3 weeks after surgery
  Objective response referred to participants with complete response (CR) or partial response (PR). CR: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: greater than or equal to (>=) 30% decrease in sum of the longest diameter (LD) of all target lesions taking as reference the screening sum LD. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments that should have been performed no less than 4 weeks after the criteria for response were first met. Longer intervals as determined by the study protocol were also appropriate. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Percentage of Participants With Clinically Significant Improvement in European Organisation for Research and Treatment of Cancer Quality of Life Core Module 30 (EORTC Quality of Life Questionnaire (QLQ)-C30) Score | Day 1 of each treatment cycle, at the study drug completion visit, and thereafter at follow-up
  The EORTC QLQ-C30 is a validated, cancer-specific 30-item patient-reported measure, and contains 14 domains to assess the impact of cancer treatment on 5 aspects of participants functioning (physical, role, cognitive, emotional, and social), 9 aspects of disease/treatment-related symptoms (fatigue, nausea and vomiting, pain, dyspnea, insomnia, loss of appetite, constipation, diarrhea) and a global QoL/overall health status scale. Questions used 4 point scale (1 'Not at all' to 4 'Very much'; with the exception of the QoL/health status scale which uses a 7-point scale (1 'very poor' to 7 'Excellent'). Each scale is transformed on a scale of 0-100; a higher score equals (=) a better level of functioning or greater degree of symptoms. Change of greater than or equal to (>=) 10-points has been found to be clinically significant. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Adverse events | 3 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Principal Investigator — Hebei Medical University Fourth Hospital; Jun Wang, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China